CLINICAL TRIAL: NCT03318068
Title: A Feasibility Study Examining the Impact of Out-patient Yoga on Children Receiving Chemotherapy
Brief Title: Outpatient Yoga Study for Adolescents Receiving Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Pediatric Oncology Group of Ontario (Other)
Responsible Party: Principal Investigator, Lillian Sung, Pediatric Oncologist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: REB# 1000054681
Record Dates: First submitted 2017-04-11; First posted 2017-10-23 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Pediatric Cancer; Quality of Life; Cancer, Treatment-Related; Psychological Distress; Yoga; Feasibility
Keywords: Cancer; Pediatric cancer; Yoga; Psychological distress; Outpatient chemotherapy
MeSH Terms: conditions — Neoplasms; Neoplasms, Second Primary

STUDY DESIGN:
Intervention Model Description: This is a feasibility study to determine if a yoga intervention can be delivered via to outpatients receiving chemotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yoga intervention arm (Experimental): The group will receive a weekly yoga session for the duration of 10 weeks. The yoga sessions will be delivered in person for 3 weeks during the intervention, coordinated with existing clinic visits. The other 7 sessions will be delivered via skype. The participant will be asked to fill out questionnaires during each of the three in-person yoga visits asking about psychological symptoms and quality of life.
  Interventions: Other: Yoga Intervention

INTERVENTIONS:
Other: Yoga Intervention — The yoga intervention will consist of a combination of yoga postures, gentle stretches, breathing techniques and relaxation. The sessions will be delivered one-on-one and will be adapted to accommodate the patients each day.

SUMMARY:
LAY SUMMARY:

The diagnosis and treatment of pediatric cancer is a significant stressor for adolescents and their families . Although most adolescents cope well with their cancer diagnosis, many experience emotional distress. A small proportion of those diagnosed with cancer will experience more intense mental distress, such as depression, anxiety, or anger. The practice of yoga may be a possible way of treating the negative emotional symptoms experienced by these adolescents. Previous studies suggest that yoga may improve anxiety, mood and psychological distress in adults with cancer. The results of two recent pediatric pilot studies show that yoga programs improved quality of life for adolescents receiving cancer treatment. Given this, we wish to examine the feasibility of offering a 10-week yoga program for adolescents who are receiving outpatient chemotherapy. This program includes both one-on-one in-person sessions and home-based sessions offered using SkypeTM. To assess this program, we will monitor patients' attendance, ask their opinions of the program and evaluate whether yoga improved their mental well-being. This study represents an important step toward identifying possible treatments to improve patients' quality of life and emotional health.

DETAILED DESCRIPTION:
Background: The diagnosis and treatment of pediatric cancer is often a distressing time for patients and families. Moreover, a subset of patients experience significant negative psychological symptoms at time of diagnosis. Often times, these symptoms persist throughout treatment, and, possibly, for years after their diagnosis. Available evidence suggests that early identification and intervention for these psychological symptoms may reduce their short-term and long-term impact. Yoga has emerged as a potential therapeutic intervention to improve psychosocial wellness with promising preliminary results in adult cancer populations.

Objective: To determine the feasibility of a 10-week, weekly yoga intervention for adolescents with cancer currently receiving cancer therapy.

Methods: This pilot study will consist of 45-minute yoga sessions administered weekly for 10 (+/- 2) consecutive weeks. Three sessions will take place in-person, timed in conjunction with participants' clinic appointments, with the remainder of sessions administered at home, through SkypeTM. Each session will be one-to-one and conducted by a yoga instructor. Participants will also complete home exercises in between these weekly sessions. Adolescents ages 10 to 18 with any cancer diagnosis will be eligible for this study. Feasibility, the primary objective, will be determined by 1) the number of patients who are recruited for this study, and 2) the number of patients who in attend at least 60% of administered sessions. The feasibility, acceptability and utility of measuring participants' emotional distress and quality of life will be examined as secondary outcomes. These outcomes will be measured at baseline, mid-way and at the end of the intervention. The Patient Reported Outcomes Measurement Information System measures for anxiety, depression and anger will be used to measure emotional distress. Patient's fatigue and quality of life will be determined using the Pediatric Quality of Life Inventory Fatigue and Acute Cancer Modules. Study enrollment is planned at 10 participants, as this sample size will enable to assess if our intervention and measurements tool are appropriate.

Significance: This study represents an important first step in determining if yoga programs can be offered at home, and if such programs influence patient well-being. If feasible, outpatient yoga programs may offer a practical and cost-effective tool to provide enhanced psychosocial wellbeing among adolescents undergoing cancer therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 10 to 18
* Receiving active cancer therapy within 21 days of enrollment and for the 10 weeks of the study
* Able to perform yoga at home (the yoga is modified at home so that it low impact exercises and fit the capabilities of the patient)
* Planned to be outpatients for more than 75 % of study

Exclusion Criteria:

* Sarcoma patients with future planned surgical interventions (can be enrolled after surgery)
* Planned HSCT during the 10 week study period

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-02-13 (Actual); Study Completion 2018-02-13 (Actual)

PRIMARY OUTCOMES:
Feasibility of delivering weekly yoga sessions to outpatients receiving chemotherapy. | Intervention runs for 10 weeks, and is administered one-on-one; study will be enrolling for 1 year with a goal to enroll 10 participants on this study. We will determine feasibility once all 10 participants have completed the study after 1 year.
  Will be determined by both the number of patients who are recruited for this study, and the number of patients who attend at least 60% of administered sessions. We will aim to enroll 10 participants at SickKids over one year. Compliance will be defined as the number of participants who complete 6 (60%) of the scheduled yoga sessions. Feasibility will be met if at least 80% (8) of participants meet this threshold of participation.

SECONDARY OUTCOMES:
Pediatric Quality of Life (PedsQL) Multidimensional Fatigue Scale Acute Version, Version 3.0 | Measure will be completed at three timepoints: 1) week 1, 2) week 4, 5 or 6 (coordinated with their medical clinic appointments), and 3) at week 10 (upon completion of the study). A change score will be used to assess changes in fatigue from week 1- 10.
  Measures self-reported fatigue; 5-point likert scale ranging from 0(almost never) to 4 (almost always), with higher scores indicating higher problems; there is no weighting of items. Scores are transformed on a scale from 0 to 100.Items are reversed scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. Mean score is calculated= Sum of the items over the number of items answered.
  Total Score is used and calculated by: Sum of all the items over the number of items answered on all the Scales. Higher scores indicate lower problems.
Pediatric Quality of Life (Peds QL) Cancer Module Acute Version | Measure will be completed at three timepoints: 1) week 1, 2) week 4, 5 or 6 (coordinated with their medical clinic appointments), and 3) at week 10 (upon completion of the study). A change score will be used to assess changes in symptoms from week 1- 10.
  Measures self-reported symptoms related to cancer treatment, capturing physical, psychological and cognitive health. 5-point likert scale ranging from 0(almost never) to 4 (almost always); there is no weighting of items. Scores are transformed on a scale from 0 to 100. Items are reversed scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. Mean score is calculated= Sum of the items over the number of items answered.
  Total Score is used and calculated by: Sum of all the items over the number of items answered on all the Scales. Higher scores indicate lower problems.
Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Anxiety Short Form 8b | Measure will be completed at three timepoints: 1) week 1, 2) week 4, 5 or 6 (coordinated with their medical clinic appointments), and 3) at week 10 (upon completion of the study). A change score will be used to assess changes in anxiety from week 1- 10.
  The PROMIS Anxiety instruments measure self-reported fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), and somatic symptoms related to arousal (racing heart, dizziness). 5-point Likert scale ranging from 1 (never) to 5 (almost always); there are 8 questions in this measure. First a raw total score is calculated by added up the values to each question, ranging from 5-40. The total raw score is then converted into a T-score using the conversion table. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 1. A higher PROMIS T-score represents more of the concept being measured, in this case, anxiety symptoms.
Patient-Reported Outcomes Measurement Information System (PROMIS) Anger - Fixed Form | Measure will be completed at three timepoints: 1) week 1, 2) week 4, 5 or 6 (coordinated with their medical clinic appointments), and 3) at week 10 (upon completion of the study). A change score will be used to assess changes in anger from week 1- 10.
  The PROMIS Anger instruments measure self-reported angry mood (irritability, frustration), negative social cognitions (interpersonal sensitivity, envy, disagreeableness), and efforts to control anger. This measure includes 5 questions. 5-point Likert scale ranging from 1 (never) to 5 (almost always) First a raw total score is calculated by added up the values to each question, ranging from 5-25. The total raw score is then converted into a T-score using the conversion table. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 1. A higher PROMIS T-score represents more of the concept being measured, in this case, anger.
Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Depressive Symptoms- Short Form 8a | Measure will be completed at three timepoints: 1) week 1, 2) week 4, 5 or 6 (coordinated with their medical clinic appointments), and 3) at week 10 (upon completion of the study). A change score will be used to assess changes in mood from week 1- 10.
  The PROMIS Depression instruments assess self-reported negative mood (sadness, guilt), views of self (selfcriticism, worthlessness), and social cognition (loneliness, interpersonal alienation), as well as decreased positive affect and engagement (loss of interest, meaning, and purpose). Somatic symptoms (changes in appetite, sleeping patterns) are not included. The Depression short form is universal rather than disease-specific. This measure includes 8 questions. 5-point Likert scale ranging from 1 (never) to 5 (almost always). It assesses depression over the past seven days. First a raw total score is calculated by added up the values to each question, ranging from 5-40. The total raw score is then converted into a T-score using the conversion table. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 1. A higher PROMIS T-score represents more of the concept being measured, in this case, depression symptoms.
Symptom Screening in Pediatrics (SSPedi) | Intervention runs for 10 weeks; Measure will be completed at three timepoints throughout the study: 1) week 1, 2) week 4, 5 or 6 (coordinated with their medical clinic appointments), and 3) at week 10 (upon completion of the study)
  Self-reported symptom screening questionnaire asking pediatric patients (age 8-18) how bothered they are by 15 identified symptoms and side effects of cancer treatment. This 5-point Likert scale score from 0 (not bothered at all) to 4 (extremely bothered), and has a total score ranging from 0-60, with a higher number indicating more bother cancer-related symptoms. Likert scores will be summed for a total score that ranges from 0 (none) to 60 (worst possible).
Acceptability of the yoga program | At the final assessement timepoint, at week 10 for each participant.
  Acceptability of the yoga program will be measured using a 5-point Likert scale at week 10. At each assessment point (week 1, week4, 5, or 6 and week 10), participants will be interviewed using open-ended questions to assess their views of the program. Likert items score from 1(strongly agree) to 5(strongly disagree) a higher score indicating greater acceptability of the yoga program.
Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Fatigue- Short Form | Measure will be completed at three timepoints: 1) week 1, 2) week 4, 5 or 6 (coordinated with their medical clinic appointments), and 3) at week 10 (upon completion of the study). A change score will be used to assess changes in fatigue from week 1- 10.
  The PROMIS Fatigue instruments evaluate a range of self-reported symptoms. Fatigue is divided into the experience of fatigue (frequency, duration, and intensity) and the impact of fatigue on physical, mental, and social activities. The Fatigue short form is universal rather than disease-specific. It assesses fatigue over the past seven days This measure includes 10 questions. 5-point Likert scale ranging from 1 (never) to 5 (almost always).First a raw total score is calculated by added up the values to each question, ranging from 5-50. The total raw score is then converted into a T-score using the conversion table. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 1. A higher PROMIS T-score represents more of the concept being measured, in this case, depression symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Sung, MD, PhD, Principal Investigator — Pediatric Oncologist, Senior Scientist
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stein E, Rayar M, Krishnadev U, Gupta A, Hyslop S, Plenert E, Schechter-Finkelstein T, Sung L. A feasibility study examining the impact of yoga on psychosocial health and symptoms in pediatric outpatients receiving chemotherapy. Support Care Cancer. 2019 Oct;27(10):3769-3776. doi: 10.1007/s00520-019-04673-9. Epub 2019 Feb 2. PMID 30712097